CLINICAL TRIAL: NCT05042427
Title: Psychometric Properties of Pregnancy Weight Management Health Literacy Questionnaire
Brief Title: Pregnancy Weight Management Health Literacy Questionnaire
Acronym: PWMHLQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chao-Hui, Lee (Other)
Collaborators: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Chao-Hui, Lee, Head Nurse of Obstetrics and Gynecology Department, Shin Kong Wu Ho-Su Memorial Hospital
Organization: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Other Study IDs: 20201209R
Record Dates: First submitted 2021-08-17; First posted 2021-09-13 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Gestational Age and Weight Conditions; Health Knowledge, Attitudes, Practice
Keywords: primigravida women; weight management; health literacy
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primigravida women: Weight management health literacy of primigravida women.
  Interventions: Other: Pregnancy Weight Management Health Literacy Questionnaire

INTERVENTIONS:
Other: Pregnancy Weight Management Health Literacy Questionnaire — Give questionnaires to check the weight management health literacy level of primigravida women.

SUMMARY:
Worldwide obesity has continued to increase over the past decades. Among the adult women, the overweight and obesity rates in Taiwan are much higher than that of women in nearby Asian countries. In particular, the body mass index of women with low health literacy exceeds the normal range before pregnancy. Without proper supervision, the increase in body weight during pregnancy may result in multiple maternal complications, affect the newborn's health, and increase unnecessary medical expenses in Taiwan's health care system. Thus, assessing pregnant women' s health literacy to manage their body weight is of importance. However, currently, there is no appropriate instrument available in Taiwan to assist health practitioners in assessing the health literacy of pregnant women for weight management. The aim of the study is to develop an instrument to measure the health literacy regarding weight management of pregnant women and examine its psychometric properties.

DETAILED DESCRIPTION:
This study will use a multiphase prospective longitudinal design. While developing the items of the instrument based on the review of the literature, five content experts will be invited to participate in the study for examining the appropriateness of the generated items. Upon the approval of the Institutional Review Board, a convenience sample will be recruited to establish face validity. Then the instrument will be refined according to the report derived from the pretesting. The content experts will then review the revised instrument again, and another 330 primigravida women will be enrolled in the study for assessing the psychometric properties. The validity and reliability of the instrument will be examined through evaluating the internal consistency reliability, split-half reliability, concurrent validity, and predictive validity. Health practitioners can use this newly developed instrument to assess pregnant women's health literacy to help manage their weight gain during pregnancy. By utilizing this instrument, health practitioners can provide individually tailored nursing care to improve the effectiveness of their weight management.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida women
* Fluent in writing, reading and speaking Mandarin

Exclusion Criteria:

* Non-pregnant
* Can't fluent in writing, reading and speaking Mandarin
* Cognitive dysfunction

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primigravida women
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
weight management health literacy | during pregnancy(before delivery/ Within 10 months)
  level of maternal weight management health literacy

SECONDARY OUTCOMES:
postpartum body weight | On the day of delivery
  record postpartum body weight in kilograms
body weight before pregnancy | On the day of delivery
  record body weight in kilograms from medical records
time of labor | On the day of delivery
  record time of labor from medical records
labor conditions | On the day of delivery
  record conditions of labor from medical records
newborn body weight | On the day of delivery
  record newborn body weight in grams from medical records
newborn body height | On the day of delivery
  record newborn body height in meters from medical records
newborn Apgar score | On the day of delivery
  record newborn Apgar score from medical records
newborn conditions | On the day of delivery
  record newborn conditions from medical records

OTHER OUTCOMES:
The short-form health literacy questionnaire (HL-SF12) | during pregnancy(before delivery/ Within 10 months)
  This study uses the short-form health literacy questionnaire (HL-SF12) to check the level of health literacy.The perceived difficulty of each health-related task was rated on 4-point Likert scales (1=very difficult, 2=difficult, 3=easy, and 4=very easy).An index value was thus obtained in which 0 represented the lowest HL and 50 the highest HL.The HL matrix was constructed from 4 steps of information processing in three health domains, which created a total of 12 dimensions or components of HL. The indices for HL were standardized to unified metrics from 0 to 50 using the formula; Index=(mean-1)×(50/3), where Index is the specific index calculated, mean is the mean of all participating items for each individual, 1 is the minimal possible value of the mean (leading to a minimum value of the index of 0), 3 is the range of the mean, and 50 is the chosen maximum value of the new metric.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yi Tai, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duong VT, Lin IF, Sorensen K, Pelikan JM, Van Den Broucke S, Lin YC, Chang PW. Health Literacy in Taiwan: A Population-Based Study. Asia Pac J Public Health. 2015 Nov;27(8):871-80. doi: 10.1177/1010539515607962. Epub 2015 Sep 29. PMID 26419635
- [Background] Huang YJ, Lin GH, Lu WS, Tam KW, Chen C, Hou WH, Hsieh CL. Validation of the European Health Literacy Survey Questionnaire in Women With Breast Cancer. Cancer Nurs. 2018 Mar/Apr;41(2):E40-E48. doi: 10.1097/NCC.0000000000000475. PMID 28221213
- [Background] Sorensen K, Van den Broucke S, Pelikan JM, Fullam J, Doyle G, Slonska Z, Kondilis B, Stoffels V, Osborne RH, Brand H; HLS-EU Consortium. Measuring health literacy in populations: illuminating the design and development process of the European Health Literacy Survey Questionnaire (HLS-EU-Q). BMC Public Health. 2013 Oct 10;13:948. doi: 10.1186/1471-2458-13-948. PMID 24112855
- [Background] Duong TV, Aringazina A, Kayupova G, Nurjanah, Pham TV, Pham KM, Truong TQ, Nguyen KT, Oo WM, Su TT, Majid HA, Sorensen K, Lin IF, Chang Y, Yang SH, Chang PWS. Development and Validation of a New Short-Form Health Literacy Instrument (HLS-SF12) for the General Public in Six Asian Countries. Health Lit Res Pract. 2019 Apr 10;3(2):e91-e102. doi: 10.3928/24748307-20190225-01. eCollection 2019 Apr. PMID 31294310
- [Background] Duong TV, Nguyen TTP, Pham KM, Nguyen KT, Giap MH, Tran TDX, Nguyen CX, Yang SH, Su CT. Validation of the Short-Form Health Literacy Questionnaire (HLS-SF12) and Its Determinants among People Living in Rural Areas in Vietnam. Int J Environ Res Public Health. 2019 Sep 11;16(18):3346. doi: 10.3390/ijerph16183346. PMID 31514271